CLINICAL TRIAL: NCT01323426
Title: Autologous Muscle Fiber Transplantation for Repair of the Urethral Sphincter in Patients With Stress Urinary Incontinence
Brief Title: Treatment of Stress Urinary Incontinence by Injection of Autologous Muscle Fibers Into the Urethral Sphincter.
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Copenhagen University Hospital at Herlev (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-1-2009-079 and H-1-2011-032
Record Dates: First submitted 2011-03-21; First posted 2011-03-25 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Urinary Incontinence, Stress
Keywords: urinary incontinence, stress; autologous
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- periurethral injection (Experimental): Periurethral injection of autologous muscle fibers
  Interventions: Procedure: Periurethral injection

INTERVENTIONS:
Procedure: Periurethral injection — Periurethral injection of autologous muscle fibers

SUMMARY:
This pilot study examines safety and efficacy of a simple procedure for treatment of stress urinary incontinence. A muscle biopsy is taken from the thigh, minced and injected into the urethral sphincter.

ELIGIBILITY:
Inclusion Criteria:

* Stress urinary incontinence refractory to conservative treatment.

Exclusion Criteria:

* urge urinary incontinence
* Pregnancy
* Pelvic organ prolapse > grade 1

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-05; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Frequency of incontinence episodes | 12 months
  Reduction in the number of leakages in three days

SECONDARY OUTCOMES:
International Consultation on Incontinence (ICIQ)short form incontinence score | 12 months
Intraurethral pressure measured by reflectometry | 12 months
Uroflow | 12 months
Adverse events peri- or postoperatively | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Søren Gräs, MD, Principal Investigator — Herlev Hospital
Locations (1):
- Herlev Hospital, Herlev, Denmark